CLINICAL TRIAL: NCT01880658
Title: Phase II Clinical Trial: Capecitabine Maintenance Therapy in Colorectal Cancer Patients With Stage IIIC and R0-R1 Resected Stage IV
Brief Title: Phase II Study of Maintenance Capecitabine to Treat Resectable Colorectal Cancer
Acronym: CAMCO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, associate professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU03
Record Dates: First submitted 2013-06-05; First posted 2013-06-19 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Neoplasms
Keywords: Maintenance therapy; Capecitabine; Adjuvant chemotherapy; Post-operation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Patients undergo R0-R1 resection and receive adjuvant chemotherapy FOLFOX or Capox for no less than 4 months. Radiotherapy may be applied for patients with rectal cancer if clinicians suspect that is necessary. Then patients receive oral capecitabine for 12 months maintenance.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000mg/m2,po(orally) on day 1-14 of 21 day cycle. Number of cycles: 16 cycles (1 year)
  Other Names: Xeloda

SUMMARY:
RATIONALE: Surgical resection and adjuvant therapy has become the main treatment for resectable colorectal cancer. Treatment with current strategies, however,recurrent rate is high for stage IIIC or R0 resected stage IV. The efficacy and safety of maintenance therapy with capecitabine is still unknown.

PURPOSE: This single arm study is exploring surgical resection and adjuvant chemotherapy followed by maintenance therapy with capecitabine to see the efficacy and safety, then to investigate the effect of maintenance therapy for stage IIIC or R0 resected stage IV colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES Primary evaluate the disease free survival rate of three years in patients with stage IIIC or resectable stage IV colorectal cancer treated with maintenance capecitabine.

Secondary

1. Evaluate the over all survival time in patients treated with these regimens.
2. Correlate genetic patterns and the presence or absence of specific tissue biomarkers with response and prognosis in patients treated with these regimens.
3. Determine quality of life (QOL) of patients treated with maintenance capecitabine versus chemotherapy termination.
4. Determine the toxic effects of maintenance regimens in these patients.
5. Determine the convenience of care in patients treated with maintenance regimens.

OUTLINE: This is a single arm, single-enter study. Patients are receiving therapies as below.

Patients undergo R0-R1 resection and receive adjuvant chemotherapy oxaliplatin with fluorouracil (5FU) and folinic acid（FOLFOX）or oxaliplatin with oxaliplatin with capecitabine(capox) for no less than 4 months. Radiotherapy may be applied for patients with rectal cancer if clinicians suspect that is necessary. Then patients receive oral capecitabine for 12 months maintenance.

Quality of life is assessed at completion of adjuvant treatment, at completion of maintenance chemotherapy , and at 1 year after maintenance chemotherapy.

After completion of adjuvant treatment, patients are followed every 3 months for 2 years, and then every 6 months for 3years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 3 years.

Eligibility Ages Eligible for Study: 18-80 Years old Genders Eligible for Study: Both Accepts Healthy Volunteers: No

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Adenocarcinoma of the colon or rectum
2. Age:18-80 years old
3. Received curative resection when diagnosed as colorectal cancer, postoperative stage: IIIC OR IV(R0 resected)
4. Adjuvant chemotherapy with mFOLFOX6 or XELOX for more than four months 5.15 days prior recruit, meet the following criteria:

   * Hematopoietic
   * Absolute neutrophil count ≥ 1,500/mm^3
   * Platelet count ≥ 100,000/mm^3
   * Hepatic
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Alkaline phosphatase ≤ 2 times ULN
   * Aspartate transaminase ≤ 2.5 times ULN
   * Alanine transaminase ≤ 2.5 times ULN
   * No hepatic disease that would preclude study treatment or follow-up
   * No uncontrolled coagulopathy
   * Renal
   * Creatinine clearance > 50 mL/min
   * No renal disease that would preclude study treatment or follow-up

6.The ECOG scores: 0～1

Exclusion Criteria:

1. Other colorectal cancers (i.e.sarcoma,lymphoma,carcinoid,squamous cell carcinoma,or cloacogenic carcinoma)
2. Synchronous cancer of other site
3. Hypersensitivity to capecitabine
4. No More than 4 weeks since prior participation in any investigational drug study
5. Clear indication of involvement of the pelvic side walls by imaging With distant metastasis
6. History of invasive rectal malignancy, regardless of disease-free interval Fertile patients must use effective contraception
7. Uncontrolled hypertension
8. Cardiovascular disease that would preclude study treatment or follow-up
9. Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
10. Pregnant or nursing, Fertile patients do not use effective contraception
11. Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
12. No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival rate(DFS) | 36 months
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Over all survival,genetic patterns, quality of life, toxic effects, convenience | 5 years
  1. Evaluate the over all survival time in patients treated with these regimens.
  2. Correlate genetic patterns and the presence or absence of specific tissue biomarkers with response and prognosis in patients treated with these regimens.
  3. Determine quality of life (QOL) of patients treated with maintenance capecitabine versus chemotherapy termination.
  4. Determine the toxic effects of maintenance regimens in these patients.
  5. Determine the convenience of care in patients treated with maintenance regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ling J, Lin Z, Shi L, Lin Y, Liu X, Lin J, Li J, Zhang J, Hu H, Cai Y, Deng Y. Capecitabine maintenance therapy in metastatic colorectal cancer patients with no evidence of disease: CAMCO trial. Future Oncol. 2023 Sep;19(30):2045-2054. doi: 10.2217/fon-2023-0149. Epub 2023 Oct 10. PMID 37814832